CLINICAL TRIAL: NCT06361940
Title: Molecular Analyses to Predict Pathways of Endocrine Resistance Following Short Term Neoadjuvant Endocrine Treatment in Patients With Hormone Receptor-Positive HER2-negative Breast Cancer (MAPPER)
Brief Title: Molecular Analyses to Predict Pathways of Endocrine Resistance Following Short Term Neoadjuvant Endocrine Treatment in Patients With Hormone Receptor-Positive HER2-negative Breast Cancer
Acronym: MAPPER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Lubna Chaudhary, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00052561
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: hormone receptor-positive; HER2-negative; endocrine therapy; neoadjuvant; anastrozole; letrozole; exemestane; tamoxifen
MeSH Terms: conditions — Breast Neoplasms | interventions — Aromatase Inhibitors; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard-of-care Endocrine therapy (Experimental): Once enrolled, patients would be treated with the current standard-of-care endocrine therapy.
  Interventions: Drug: Aromatase inhibitors or tamoxifen

INTERVENTIONS:
Drug: Aromatase inhibitors or tamoxifen — Choice of endocrine therapy (aromatase inhibitors or tamoxifen) would be decided by medical oncologist, following a review of the patient's medical history and menstrual status.

SUMMARY:
This is an exploratory phase II interventional study that initiates standard-of-care anti-estrogen treatment preoperatively for 4-12 weeks (+/- 2 weeks).

DETAILED DESCRIPTION:
Patients with HR+ HER2- node-negative breast cancers generally undergo surgical resection upfront, followed by adjuvant chemotherapy, if needed, in addition to adjuvant endocrine therapy. Because endocrine therapy is primarily delivered in the postoperative setting, the ability to assess the tumor response to this treatment modality is lost and very difficult to assess. This study offers the unique opportunity to assess the responsiveness of breast tumors to endocrine therapy while the tumors are still in vivo by treating patients with endocrine therapy before surgery and assessing molecular changes with treatment. By comparing pre- and post-treatment levels of molecular markers with advanced omic analysis in individual tumors, the investigators expect to identify predictors of responsiveness to existing agents and identify new candidate therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral diagnostic breast mammogram and ultrasound within 60 days of enrollment.
2. Pathologically proven diagnosis of invasive breast cancer, clinical stage I or II.
3. Patients must be clinically lymph node negative. Lymph node negativity must be confirmed by clinical exam and/or ultrasound imaging.
4. The patient must be female.
5. Age ≥18 years.
6. Estrogen and/or progesterone receptor positive tumor defined ≥1% positively staining cells by immunohistochemistry, according to the current American Society of Clinical Oncology/College of American Pathologists guidelines.
7. Human epidermal growth factor receptor 2 (HER2) /neu must be negative by immunohistochemistry (IHC) or fluorescence in situ hybridization (FISH).
8. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
9. Bilateral breast cancer and/or multifocal, multicentric disease is allowed.
10. Appropriate pretreatment evaluations for protocol entry, including no clinical evidence for distant metastases, based upon the following minimum diagnostic workup: history/physical examination, including breast exam (inspection and palpation of the breasts), clinically negative axillary lymph nodes, within 28 days prior to study entry.
11. The patient must qualify for endocrine treatment (treatment of choice), per the treating medical oncologist.
12. The patient must provide study-specific informed consent prior to study entry.
13. Patients with a prior history of breast cancer will be considered eligible, if they have completed all treatment (including endocrine therapy) more than two years prior to registration.
14. Patients must not have had a prior treatment for this breast cancer or for any malignancy diagnosed or treated within the past two years, with the exception of non-melanomatous skin cancer, carcinoma in situ of the cervix.
15. Women of childbearing age will be advised to use adequate methods of contraception. Adequate methods of contraception for premenopausal women include barrier methods and/or non-hormonal methods (Intrauterine devices etc.).
16. Strong cytochrome P450 2D6 (CYP2D6) inhibitors will be prohibited with tamoxifen, as it can decrease the efficacy of tamoxifen. There are no known strong interactions with aromatase inhibitors.

Exclusion Criteria:

1. American Joint Committee on Cancer (AJCC) clinical T4, N1-3 or M1, breast cancer.
2. Synchronous non-breast malignancy (exceptions include non-melanomatous skin cancer, carcinoma in situ of the cervix).
3. Purely noninvasive breast cancer (i.e., ductal carcinoma in situ, lobular carcinoma in situ).
4. Men with breast cancer. Male breast cancer is a rare event and it is unclear if neoadjuvant endocrine treatment approach is safe in men.
5. Medical, psychiatric or other condition that would prevent the patient from receiving the protocol therapy or providing informed consent.
6. Pregnant or lactating women are ineligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the number of subjects with increased HER-1 receptor tyrosine kinases protein expression in tumors. | Time of surgery
  Pathologists will use immunohistochemistry (IHC) to determine the average count of tumor protein expression. IHC is reported categorically as 0,1, 2 or 3. Any increase between these categories is considered increase.
Change from baseline in the number of subjects with increased HER-2 receptor tyrosine kinases protein expression in tumors. | Time of surgery
  Pathologists will use immunohistochemistry to determine the average count of tumor protein expression. IHC is reported categorically as 0,1,2 or 3. Any increase between these categories is considered increase.
Change from baseline in the number of subjects with increased HER-3 receptor tyrosine kinases protein expression in tumors. | Time of surgery
  Pathologists will use immunohistochemistry to determine the average count of tumor protein expression. IHC is reported categorically as 0,1,2 or 3. Any increase between these categories is considered increase.
Change from baseline in the number of subjects with increased HER-4 receptor tyrosine kinases protein expression in tumors. | Time of surgery
  Pathologists will use immunohistochemistry to determine the average count of tumor protein expression. IHC is reported categorically as 0,1,2 or 3. Any increase between these categories is considered increase.

CONTACTS AND LOCATIONS:
Overall Officials: Lubna N Chaudhary, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No